CLINICAL TRIAL: NCT06260514
Title: A Phase 1, Open-Label, Multicenter, First-In-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of APR-1051 in Patients With Advanced Solid Tumors
Brief Title: Study of APR-1051 in Patients With Advanced Solid Tumors
Acronym: ACESOT-1051
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APR-1051-001
Record Dates: First submitted 2024-01-18; First posted 2024-02-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APR-1051 (Experimental): Dose Escalation based on BOIN Design
  Interventions: Drug: APR-1051

INTERVENTIONS:
Drug: APR-1051 — WEE1 Inhibitor

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of APR-1051 through the performance of a Phase 1, open-label, safety, PK, and preliminary efficacy study of oral APR-1051 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of advanced/metastatic solid tumor
* Measurable or evaluable disease per RECIST version 1.1 (radiographic disease progression per PCWG3 criteria for patients with mCRPC)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 or Karnofsky Performance Status (KPS) ≥ 70%
* Patients must have recovered to Grade 1 or baseline levels from toxicity or adverse events related to prior treatment for their cancer, excluding Grade ≤ 2 neuropathy, alopecia, or skin pigmentation
* Adequate bone marrow and organ function
* Women of child-bearing potential (WOCBP) or men of child-fathering potential must agree to use adequate contraception prior to study entry

Exclusion Criteria:

* Patient has had prior systemic anti-cancer therapy (cytotoxic chemotherapy, immunotherapy, targeted therapy) within 3 weeks (6 weeks in cases of mitomycin C, nitrosourea, lomustine) or at least 5 half-lives (whichever is shorter, but no less than 2 weeks) prior to Day 1
* Prior radiation therapy at the target lesion unless there is evidence of disease progression. If patient has had prior radiation therapy for disease progression, see Exclusion Criterion 1 for allowed interval between radiotherapy and Day 1 and recovery of AEs
* Treatment with any investigational agent administered within 30 days or 5 half-lives, whichever is shorter, before the first dose of APR-1051
* Major surgery within 21 days prior to Day 1
* Concomitant treatment with other anti-cancer therapy, including chemotherapy, immunotherapy, biological therapy, radiation therapy (except palliative local radiation therapy), or other novel anti-cancer agents. Note: endocrine therapy for breast and prostate cancer is allowed along with agents to treat or prevent skeletal related events (zoledronic acid, pamidronate, denosumab)
* Subjects with active (uncontrolled, metastatic) second malignancies or requiring therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events | Day 1 to 28, each cycle is 28 days
  * Part 1 dose escalation: Incidence of adverse Events (AE), serious AEs (SAE), treatment-related AEs, AEs that would qualify as a dose-limiting toxicity (DLT), changes in clinical laboratory values, vital signs, ECG, ECHO
  * Part 1 dose escalation: Severity of adverse Events (AE), serious AEs (SAE), treatment-related AEs, and changes in clinical laboratory values, vital signs, ECG, ECHO according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0
Recommended dose of APR-1051 | Day 1 to 28, each cycle is 28 days
  •Part 1 dose escalation: Recommended Phase 2 Dose (RP2D) of APR-1051 monotherapy [Time frame: Day 1 through to start of dose expansion phase]. The RP2D of will be determined based on review of safety, tolerability, pharmacokinetics/pharmacodynamics, and preliminary efficacy data

SECONDARY OUTCOMES:
Pharmacokinetics: Cmax/Cmin of APR-1051 | Day 1 to 112
  Plasma concentration of APR-1051: maximum (Cmax), minimum (Cmin)
Pharmacokinetics: Tmax of APR-1051 | Day 1 to 112
  Time to peak plasma concentration of APR-1051 (Tmax)
Pharmacokinetics: AUC of APR-1051 | Day 1 to 112
  Area under plasma versus time curve (AUC) of APR-1051 max)
Pharmacokinetics: t1/2 of APR-1051 | Day 1 to 112
  Half-life of APR-1051 (t1/2)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - MD Anderson Cancer Center (MDACC), Houston, Texas
  - NEXT Oncology -Dallas, Irving, Texas
  - NEXT Oncology -San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No